CLINICAL TRIAL: NCT01795261
Title: Comparative Effectiveness of Congregation and Clinic Based Approaches to Prevention of Mother to Child Transmission of HIV
Brief Title: Healthy Beginning Initiative
Acronym: HBI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Nevada, Reno (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01HD075050-01 (NIH); 1R01HD075050-01 (NIH)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lifestyle counseling: Prevention of mother to child transmission of HIV
- Lifestyle counseling Male: male partners and PMTCT completion rate among HIV-infected pregnant women.

SUMMARY:
The purpose of this study is to determine if providing free laboratory test to pregnant women and their spouses at churches, in addition to laboratories or hospitals, will increase the number of pregnant women and their spouses who get screened for HIV, malaria, sickle cell trait, hemoglobin levels, syphilis, and hepatitis B. These tests are necessary to keep mothers healthy during pregnancy and lead to healthy babies. This research is taking place in 40 churches in Nigeria.

DETAILED DESCRIPTION:
We are conducting a randomized trial to evaluate the comparative effectiveness of a congregation-based Healthy Beginning Initiative (HBI) delivered by lay health advisors (Intervention Group; IG), versus a Facility Based Approach (Control Group; CG) on the HIV testing rate and PMTCT completion among 2,700 pregnant women. Four dioceses with forty churches nested in the dioceses, will be randomly assigned to either the IG (N=2; n=20) or the CG (N=2; n=20). The HBI combines a family educational game show and an integrated on-site laboratory testing in the context of a baby shower. Monthly prayer sessions for pregnant women will be used for recruitment and a baby reception following infant baptisms will be used for follow up after delivery. The primary outcome is difference in testing rate among pregnant women in IG compared to CG. The secondary outcomes are HIV testing rate among male partners and PMTCT completion among HIV-infected pregnant women. Pregnant women will complete an investigator-administered questionnaire at the baby reception to collect information on HIV testing and PMTCT completion. Data will be confirmed with Health Facilities and on-site testing data. This proposal is a collaboration among Partners for Prevention, education, Training, Treatment and Research (PeTR-Global Solutions)/AIDSRelief (our PEPFAR-funded partner in Nigeria responsible for training, HIV testing, linkage to treatment and local oversight of the project); New York University School of Medicine (program evaluation and shares oversight with PI), Board of Regents, NSHE, obo University of Nevada, Reno (provide overall oversight, data management and evaluation of program effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females 18 years and older;
* Male partners of pregnant females 18 years and older;
* Subjects must attend church at one of the participating diocese

Exclusion Criteria:

- Subjects will be excluded if they are not pregnant women or their male partners or are younger than 18 years old.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women and their male partners who are 18 years and older and attend one of the 40 churches in the Enugu state of Nigeria will be eligible to participate in the study. All participation is voluntary.
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of HIV testing rates in pregnant women and their male partners in a congregation based approach compared to a health facility based approach. | One year
  We need to have 1,313 pregnant women in each arm of the study and follow them through pregnancy and up to 6 weeks post-delivery. Since pregnant women will be recruited at different stages of pregnancy, we will need to end recruitment 5 months after the study is open to recruitment and allow time to follow last recruited pregnant women through 9 months of pregnancy and up to 6 weeks post-delivery (approximately 11 months).

SECONDARY OUTCOMES:
Associations between HIV Test and Interventions and other covariates (risk factors) at individual- and community (church)-level will also be analyzed. | one year
  Variables include age, household income, education level, previous HIV testing, last menstrual period, marital status, and employment status. HIV testing and PMTCT completion: will be assessed using a one-page investigator-administered questionnaire completed by pregnant women during the baby reception.

CONTACTS AND LOCATIONS:
Overall Officials: Echezona Ezeanolue, MD, Principal Investigator — University of Nevada, Reno
Locations (1):
- PeTR Global Solutions, Abuja, Maitama, Nigeria

REFERENCES:
- [Background] Tubiana R, Le Chenadec J, Rouzioux C, Mandelbrot L, Hamrene K, Dollfus C, Faye A, Delaugerre C, Blanche S, Warszawski J. Factors associated with mother-to-child transmission of HIV-1 despite a maternal viral load <500 copies/ml at delivery: a case-control study nested in the French perinatal cohort (EPF-ANRS CO1). Clin Infect Dis. 2010 Feb 15;50(4):585-96. doi: 10.1086/650005. PMID 20070234
- [Background] European Collaborative Study. Mother-to-child transmission of HIV infection in the era of highly active antiretroviral therapy. Clin Infect Dis. 2005 Feb 1;40(3):458-65. doi: 10.1086/427287. Epub 2005 Jan 7. PMID 15668871
- [Background] Centers for Disease Control and Prevention (CDC). Achievements in public health. Reduction in perinatal transmission of HIV infection--United States, 1985-2005. MMWR Morb Mortal Wkly Rep. 2006 Jun 2;55(21):592-7. PMID 16741495
- [Background] Turan JM, Bukusi EA, Onono M, Holzemer WL, Miller S, Cohen CR. HIV/AIDS stigma and refusal of HIV testing among pregnant women in rural Kenya: results from the MAMAS Study. AIDS Behav. 2011 Aug;15(6):1111-20. doi: 10.1007/s10461-010-9798-5. PMID 20827573
- [Background] Nunn A, Zaller N, Cornwall A, Mayer KH, Moore E, Dickman S, Beckwith C, Kwakwa H. Low perceived risk and high HIV prevalence among a predominantly African American population participating in Philadelphia's Rapid HIV testing program. AIDS Patient Care STDS. 2011 Apr;25(4):229-35. doi: 10.1089/apc.2010.0313. Epub 2011 Mar 15. PMID 21406004
- [Background] Monjok E, Smesny A, Essien EJ. HIV/AIDS-related stigma and discrimination in Nigeria: review of research studies and future directions for prevention strategies. Afr J Reprod Health. 2009 Sep;13(3):21-35. PMID 20690259
- [Background] Hardon A, Vernooij E, Bongololo-Mbera G, Cherutich P, Desclaux A, Kyaddondo D, Ky-Zerbo O, Neuman M, Wanyenze R, Obermeyer C. Women's views on consent, counseling and confidentiality in PMTCT: a mixed-methods study in four African countries. BMC Public Health. 2012 Jan 11;12:26. doi: 10.1186/1471-2458-12-26. PMID 22236097
- [Background] Franca-Martins AM, Graubard Z, Holloway GA, Van der Merwe FJ. Placental haemangioma associated with acute fetal anemia in labour. Acta Med Port. 1990 May-Jun;3(3):187-9. PMID 2220431
- [Background] Youngleson MS, Nkurunziza P, Jennings K, Arendse J, Mate KS, Barker P. Improving a mother to child HIV transmission programme through health system redesign: quality improvement, protocol adjustment and resource addition. PLoS One. 2010 Nov 9;5(11):e13891. doi: 10.1371/journal.pone.0013891. PMID 21085479
- [Background] Ekouevi DK, Stringer E, Coetzee D, Tih P, Creek T, Stinson K, Westfall AO, Welty T, Chintu N, Chi BH, Wilfert C, Shaffer N, Stringer J, Dabis F. Health facility characteristics and their relationship to coverage of PMTCT of HIV services across four African countries: the PEARL study. PLoS One. 2012;7(1):e29823. doi: 10.1371/journal.pone.0029823. Epub 2012 Jan 20. PMID 22276130
- [Background] Okunlola MA, Ayinde OA, Owonikoko KM, Omigbodun AO. Factors influencing gestational age at antenatal booking at the University College Hospital, Ibadan, Nigeria. J Obstet Gynaecol. 2006 Apr;26(3):195-7. doi: 10.1080/01443610500508220. PMID 16698622
- [Background] Adegbola O. Gestational age at antenatal booking in Lagos University Teaching Hospital (LUTH). Nig Q J Hosp Med. 2009 Jul-Sep;19(3):162-4. PMID 20836323
- [Background] Jivegard L, Holm J, Bergqvist D, Bjorck CG, Bjorkman H, Brunius U, Claes G, Hammarsten J, Jernby B, Konrad P, et al. Acute lower limb ischemia: failure of anticoagulant treatment to improve one-month results of arterial thromboembolectomy. A prospective randomized multi-center study. Surgery. 1991 May;109(5):610-6. PMID 2020905
- [Background] Johnson LF, Stinson K, Newell ML, Bland RM, Moultrie H, Davies MA, Rehle TM, Dorrington RE, Sherman GG. The contribution of maternal HIV seroconversion during late pregnancy and breastfeeding to mother-to-child transmission of HIV. J Acquir Immune Defic Syndr. 2012 Apr 1;59(4):417-25. doi: 10.1097/QAI.0b013e3182432f27. PMID 22193774
- [Derived] Ezeanolue EE, Obiefune MC, Ezeanolue CO, Ehiri JE, Osuji A, Ogidi AG, Hunt AT, Patel D, Yang W, Pharr J, Ogedegbe G. Effect of a congregation-based intervention on uptake of HIV testing and linkage to care in pregnant women in Nigeria (Baby Shower): a cluster randomised trial. Lancet Glob Health. 2015 Nov;3(11):e692-700. doi: 10.1016/S2214-109X(15)00195-3. PMID 26475016
- [Derived] Ezeanolue EE, Obiefune MC, Yang W, Obaro SK, Ezeanolue CO, Ogedegbe GG. Comparative effectiveness of congregation- versus clinic-based approach to prevention of mother-to-child HIV transmission: study protocol for a cluster randomized controlled trial. Implement Sci. 2013 Jun 8;8:62. doi: 10.1186/1748-5908-8-62. PMID 23758933